CLINICAL TRIAL: NCT05904275
Title: A Randomized Case Control Study of Pre-emptive Caudal Epidural Analgesia With Ropivacaine With and Without Dexamethasone for Lumbosacral Spine Surgery
Brief Title: Pre-emptive Caudal Epidural Analgesia With Ropivacaine With or Without Dexamethasone in Lumbosacral Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Trauma Center (Other)
Responsible Party: Principal Investigator, Dr. Jay Prakash Thakur, Assistant professor, National Trauma Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NationalTraumaCenter
Record Dates: First submitted 2023-01-27; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group RD (Experimental): Group RD - caudal epidural injection with 0.25% ropivacaine 20 ml containing dexamethasone 8 mg (0.5% Ropivacaine 10 ml + 8 mg/2 ml Dexamethasone + 8 ml NS)
  Interventions: Drug: caudal epidural injection
- Group R (Experimental): Group R- caudal epidural injection with 0.25% ropivacaine 20 ml
  Interventions: Drug: caudal epidural injection

INTERVENTIONS:
Drug: caudal epidural injection — Preoperative Ultrasound guided caudal epidural injection in lumbosacral spine surgeries for postoperative analgesia.
  Other Names: Caudal epidural injection with ropivacaine and dexamethasone

SUMMARY:
Lumbosacral spine surgeries are commonly performed under GA. Perioperative pain following spine surgeries not only contributes to significant morbidities but also hampers early mobilization. Perioperative opioids, though relieve pain but hampers consciousness, increase PONV and delays mobilization. Caudal analgesia can be effectively given preemptively to alleviate pain and facilitate early mobilization. Caudal epidural block places the needle through the sacral hiatus into the epidural space to deliver medications. It can be performed as ultrasound guided procedure with very high successful rates. Single shot caudal block with local anesthetic provides analgesia for 2-4 hours but this can be further prolonged by adding adjuvants like opioids, steroids, ketamine, alpha 2 agonists, adrenaline etc. Ropivacaine is a long-acting amide local anesthetic agent which is less lipophilic, less cardiac and central nervous system toxicity with similar duration of analgesia, has lesser motor blockade and facilitates earlier mobilization than bupivacaine. Dexamethasone is a highly potent, long acting glucocorticoid. Caudal dexamethasone prolongs the analgesic duration of the ropivacaine. The aim of this study is to evaluate the role of pre-emptive caudal epidural analgesia for postoperative pain relief in lumbosacral surgeries and to compare the effect of adding dexamethasone to ropivacaine with respect to quality of analgesia, duration of analgesia, hemodynamic effects and associated side effects.

DETAILED DESCRIPTION:
Lumbosacral spine surgeries are commonly performed under GA. Perioperative pain following spine surgeries not only contributes to significant morbidities but also hampers early mobilization. Perioperative opioids, though relieve pain but hampers consciousness, increase PONV and delays mobilization. Caudal analgesia can be effectively given preemptively to alleviate pain and facilitate early mobilization. Caudal epidural block places the needle through the sacral hiatus into the epidural space to deliver medications. It can be performed as ultrasound guided procedure with very high successful rates. Single shot caudal block with local anesthetic provides analgesia for 2-4 hours but this can be further prolonged by adding adjuvants like opioids, steroids, ketamine, alpha 2 agonists, adrenaline etc. Ropivacaine is a long-acting amide local anesthetic agent which is less lipophilic, less cardiac and central nervous system toxicity with similar duration of analgesia, has lesser motor blockade and facilitates earlier mobilization than bupivacaine. Dexamethasone is a highly potent, long acting glucocorticoid. Caudal dexamethasone prolongs the analgesic duration of the ropivacaine. The aim of this study is to evaluate the role of pre-emptive caudal epidural analgesia for postoperative pain relief in lumbosacral surgeries and to compare the effect of adding dexamethasone to ropivacaine with respect to quality of analgesia, duration of analgesia, hemodynamic effects and associated side effects.

Patients will be allocated in one of the two groups, I and II, consisting of 30 each, using a lottery based random number. A box containing 60 chits, with 30 labelled as group I and other 30 as group II, will be given to each patient and will be asked to take out 1 chit. The group allocated will be written in separate paper by an anesthesiologist, who will also prepare drugs. Decoding will be done later after completion of all data collection. The patient in Group I will be given caudal epidural injection with 0.25% ropivacaine 20 ml containing dexamethasone 8 mg (0.5% Ropivacaine 10 ml + 8 mg/2 ml Dexamethasone + 8 ml NS) and group II will be give 0.25% ropivacaine 20 ml. All the data collection will be done by another anesthesiologist, not involved in group allocation, drug preparation and administration.

At preoperative visit, all patients will be made familiar with VAS score for pain assessment and will be recorded. At operation theatre, standard American Society of Anesthesiologists (ASA) monitoring, including electrocardiography, noninvasive blood pressure, pulse oximetry and endtidal carbon dioxide, will be applied and measured. Patient's vitals will be recorded at preinduction, induction, postintubation, after caudal injection, time of incision, and at 15 min intervals till half an hour after completion of surgery. Intravenous (IV) line will be secured, and inj. Ringer Lactate (RL) 500 ml will be administered. Anesthesia will be induced with inj. Midazolam 0.04 mg/kg, inj. Fentanyl 2 mcg/kg, inj. Propofol in titrated dosages till loss of consciousness and inj. Rocuronium 0.6 mg/kg to facilitate intubation. The time of induction will be noted. After intubation and securing airway, foley's catheterization of bladder will be done and patient will be positioned in prone position for surgery in which caudal epidural injection will also be given. After painting and draping, ultrasound guided visualization of sacral hiatus will be done. In longitudinal view, using in plane technique, 22 gauge Quincke's spinal needle will be inserted below sacrococcygeal ligament. After negative aspiration of blood and CSF, epidural space will also be confirmed by injecting 3 ml of normal saline. The prepared study drugs will be injected. The time of caudal drug administration will be noted. The surgical incision will be allowed after 20 minutes of injecting drugs in both groups, to allow fixation of drugs. The time of surgical incision will be noted. Anaesthesia will be maintained on oxygen, isoflurane and intermittent boluses of muscle relaxants. Inj. Paracetamol 1 g and inj. Diclofenac 75 mg will be given intravenously, around 1 hour before anticipated completion of surgery. Neuromuscular blockade will be reversed with inj. Neostigmine 0.05 mg/kg and inj. Glycopyrrolate 0.01 mg/kg. Patients will be extubated after return of consciousness and muscle power, and will be shifted to post-operative ward. VAS score will be recorded at immediate postoperative period, 4, 8, 12 and 24 hours. All patients will be given inj. Paracetamol 1 g 8 hourly and inj. Diclofenac 75 mg 12 hourly as an intravenous infusion. If any patients have VAS ≥ 4 at any time, rescue analgesia in form of inj. Pethidine 50 mg with inj. Promethazine 25 mg will be given intramuscularly. The time to demand of first dose of supplemental (rescue) analgesic medication will be recorded. Any complications and adverse drug reactions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing lumbosacral spine surgeries by posterior approach, including discectomy, laminectomy and laminotomy with or without instrumentation
2. ASA PS I and II
3. Age 18 to 65 years

Exclusion Criteria:

1. Patients with hypersensitivity to ropivacaine.
2. Patients with anomalies of sacral anatomy.
3. Local site infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale score | At immediate postoperative period
  postoperative Visual Analogue Scale score
Visual Analogue Scale score | At 4 hours postoperatively
  postoperative Visual Analogue Scale score
Visual Analogue Scale score | At 8 hours postoperatively
  postoperative Visual Analogue Scale score
Visual Analogue Scale score | At 12 hours postoperatively
  postoperative Visual Analogue Scale score
Visual Analogue Scale score | At 24 hours postoperatively
  postoperative Visual Analogue Scale score
Time of rescue analgesia | 24 hours
  Time of VAS score >4 asking for rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pr Thakur, MD,FIPM, Principal Investigator — National Academy of Medical Science, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinstein JN, Lurie JD, Olson PR, Bronner KK, Fisher ES. United States' trends and regional variations in lumbar spine surgery: 1992-2003. Spine (Phila Pa 1976). 2006 Nov 1;31(23):2707-14. doi: 10.1097/01.brs.0000248132.15231.fe. PMID 17077740
- [Background] Meng T, Zhong Z, Meng L. Impact of spinal anaesthesia vs. general anaesthesia on peri-operative outcome in lumbar spine surgery: a systematic review and meta-analysis of randomised, controlled trials. Anaesthesia. 2017 Mar;72(3):391-401. doi: 10.1111/anae.13702. Epub 2016 Oct 22. PMID 27770448
- [Background] Kao SC, Lin CS. Caudal Epidural Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:9217145. doi: 10.1155/2017/9217145. Epub 2017 Feb 26. PMID 28337460
- [Background] Klocke R, Jenkinson T, Glew D. Sonographically guided caudal epidural steroid injections. J Ultrasound Med. 2003 Nov;22(11):1229-32. doi: 10.7863/jum.2003.22.11.1229. PMID 14620894
- [Background] Chen CP, Wong AM, Hsu CC, Tsai WC, Chang CN, Lin SC, Huang YC, Chang CH, Tang SF. Ultrasound as a screening tool for proceeding with caudal epidural injections. Arch Phys Med Rehabil. 2010 Mar;91(3):358-63. doi: 10.1016/j.apmr.2009.11.019. PMID 20298824
- [Background] Nikooseresht M, Hashemi M, Mohajerani SA, Shahandeh F, Agah M. Ultrasound as a screening tool for performing caudal epidural injections. Iran J Radiol. 2014 May;11(2):e13262. doi: 10.5812/iranjradiol.13262. Epub 2014 May 15. PMID 25035698
- [Background] Chen CP, Tang SF, Hsu TC, Tsai WC, Liu HP, Chen MJ, Date E, Lew HL. Ultrasound guidance in caudal epidural needle placement. Anesthesiology. 2004 Jul;101(1):181-4. doi: 10.1097/00000542-200407000-00028. PMID 15220789
- [Background] Blanchais A, Le Goff B, Guillot P, Berthelot JM, Glemarec J, Maugars Y. Feasibility and safety of ultrasound-guided caudal epidural glucocorticoid injections. Joint Bone Spine. 2010 Oct;77(5):440-4. doi: 10.1016/j.jbspin.2010.04.016. Epub 2010 Sep 24. PMID 20869897
- [Background] Yoon JS, Sim KH, Kim SJ, Kim WS, Koh SB, Kim BJ. The feasibility of color Doppler ultrasonography for caudal epidural steroid injection. Pain. 2005 Nov;118(1-2):210-4. doi: 10.1016/j.pain.2005.08.014. Epub 2005 Oct 4. PMID 16213088
- [Background] Aggarwal A, Aggarwal A, Harjeet, Sahni D. Morphometry of sacral hiatus and its clinical relevance in caudal epidural block. Surg Radiol Anat. 2009 Dec;31(10):793-800. doi: 10.1007/s00276-009-0529-4. Epub 2009 Jul 4. PMID 19578805
- [Background] Kiribayashi M, Inagaki Y, Nishimura Y, Yamasaki K, Takahashi S, Ueda K. Caudal blockade shortens the time to walking exercise in elderly patients following low back surgery. J Anesth. 2010 Apr;24(2):192-6. doi: 10.1007/s00540-009-0840-6. Epub 2010 Jan 19. PMID 20084409
- [Background] Kumar S, Palaniappan JM, Kishan A. Preemptive Caudal Ropivacaine: An Effective Analgesic during Degenerative Lumbar Spine Surgery. Asian Spine J. 2017 Feb;11(1):113-119. doi: 10.4184/asj.2017.11.1.113. Epub 2017 Feb 17. PMID 28243379
- [Background] Kalappa S, Sridhara RB, Kumaraswamy S. Dexmedetomidine as an Adjuvant to Pre-Emptive Caudal Epidural Ropivacaine for Lumbosacral Spine Surgeries. J Clin Diagn Res. 2016 Jan;10(1):UC22-4. doi: 10.7860/JCDR/2016/15286.7145. Epub 2016 Jan 1. PMID 26894155
- [Background] Samagh N, Pai RK, Mathews TK, Jangra K, Varma RG. Pre-emptive caudal epidural analgesia with ropivacaine for lumbosacral spine surgery: A randomized case control study. J Anaesthesiol Clin Pharmacol. 2018 Apr-Jun;34(2):237-241. doi: 10.4103/joacp.JOACP_72_17. PMID 30104836
- [Background] Rosenberg PH, Heinonen E. Differential sensitivity of A and C nerve fibres to long-acting amide local anaesthetics. Br J Anaesth. 1983 Feb;55(2):163-7. doi: 10.1093/bja/55.2.163. PMID 6830678
- [Background] Kalappa S, Sridhar RB, Nagappa S. Comparing the Efficacy of Caudal with Intravenous Dexamethasone in the Management of Pain Following Lumbosacral Spine Surgeries: A Randomized Double Blinded Controlled Study. Anesth Essays Res. 2017 Apr-Jun;11(2):416-420. doi: 10.4103/0259-1162.194581. PMID 28663633
- [Result] Baliga S, Treon K, Craig NJ. Low Back Pain: Current Surgical Approaches. Asian Spine J. 2015 Aug;9(4):645-57. doi: 10.4184/asj.2015.9.4.645. Epub 2015 Jul 28. PMID 26240729